CLINICAL TRIAL: NCT04331756
Title: Use of Tragus Pressure in Guiding Emergence From Anaesthesia- a Randomised Controlled Trial
Brief Title: Use of Tragus Pressure in Guiding Emergence From Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/00071
Record Dates: First submitted 2020-03-26; First posted 2020-04-02 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia
Keywords: Anaesthesia Emergence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guiding Emergence From Anaesthesia Without Tragus Pressure (Other): Monitoring of patients and removal of laryngeal mask airway (LMA) as per routine practice in post anaesthesia care unit (PACU)
  Interventions: Procedure: Guiding Emergence From Anaesthesia Without Tragus Pressure
- Guiding Emergence From Anaesthesia With Tragus Pressure (Experimental): Tragus pressure documentation of planes of emergence from anaesthesia - regular 3-5 minutes follow up with Tragus pressure till removal of airway device or rejection of it by patient
  Interventions: Procedure: Guiding Emergence From Anaesthesia With Tragus Pressure

INTERVENTIONS:
Procedure: Guiding Emergence From Anaesthesia With Tragus Pressure — Use of tragus pressure in guiding patients from emergence from anaesthesia post-surgery
  Arms: Guiding Emergence From Anaesthesia With Tragus Pressure
Procedure: Guiding Emergence From Anaesthesia Without Tragus Pressure — Usual clinical routine practice in guiding patients from emergence from anaesthesia post-surgery
  Arms: Guiding Emergence From Anaesthesia Without Tragus Pressure

SUMMARY:
The aims of this study is to evaluate the effectiveness of tragus pressure application in predicting or facilitating recovery from general anaesthesia, and compare the reliability of tragus pressure guided recovery/ emergence from anaesthesia to conventional modes of recovery

DETAILED DESCRIPTION:
More than 70% of general anaesthesia are now performed with laryngeal mask (LMA) as the airway support device with state of the art intra-operative monitoring such as end tidal inhalational anaesthetic agent concentration and fronto-temporal electroencephalographic waves analysis such as the Bispectral index score (BIS) and entropy. The use of LMAs have promised rapid turnover allowing more patients to be operated in the limited operating theatres' time. This comes with the additional price of losing the continuity of advanced monitoring devices in the post anaesthesia units, the best being end tidal carbon dioxide analysis. When patients are brought to the PACU, much of the monitoring of emergence from anaesthesia is fairly done through clinical measures such as motor activity, response to auditory stimuli, tactile taps on shoulder and occasional nociceptive stimuli such as sternal rub. The timing of the responsiveness of these stimuli is unknown and nursing support teams are unable to suggest a frame of time on when the patient would recover. One of the main reasons for this unpredictability is that the recovery is not planned based on the last recorded end tidal anaesthetic agent concentration before leaving the operating theatre to be shifted to PACU, but by an approximation of time since the patient has arrived in PACU and by early signs of recovery such as appearance of forehead wrinkles or motor activities. The incidence of airway events such as laryngospasm, obstruction after removal of airway devices, desaturations from resedation/ apnea and rescue measures such as reintubation/ ambu ventilation needed globally and from our local data is up to 1-5%. The incidence is higher with children and patients with reactive airways, obesity and associated complicating comorbidities. Using BIS monitoring and end tidal agent analysis for each of the 18 post anaesthesia care unit bays for recovering patients scientifically is not a cost-effective initiative. The tragus pressure technique has been known to be appropriate stimuli that has adequate stimulation of reticular activating system (RAS) without producing nociception that can trigger airway events such a laryngospasm. Physiological sleep studies have quoted that tragus pressure can contribute to arousal without causing vagotonic response that is known to occur from 'startle response' or sudden emergence. Through this study we propose to evaluate the consistency in predictability of recovery from general anaesthesia and deep sedation with Ramsay score 3 through application of tragus pressure. The presence of reflex pupillary dilatation and early signs of recovery such as swallowing, gentle grimace and minor peripheral motor movements, we propose, gives a predictable plane of recovery from anaesthesia where the LMAs are removed safely without treading the dreaded stage 2 of excitability of anaesthesia. The proposed method also allows for continued responsiveness of patient with coherent verbal responses to auditory stimuli after safe removal of the airway, thereby minimizing the incidence of airway complication and hence the interventions required for the same. The continued alert responsiveness of the patient also allows for the post anaesthesia unit team to attend to other patients who might need more immediate care.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2
* Surgeries with no risk of aspiration
* Patients with laryngeal mask airway (LMA) insitu on arrival in the PACU
* Surgery duration < 4 hours

Exclusion Criteria:

* ASA 3 and 4
* Organ failure with decompensation : Eg Heart failure, renal failure, liver failure
* History of psychiatric illness or medications for mood control
* Pregnancy
* Patients for neurosurgery or GCS <12/15
* LMA used for failed intubation or difficult airway protocol
* Patients with no LMA on arrival in the PACU
* Patients who are awake with LMA/ Responding to call on arrival at PACU

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Differences in time and ease of LMA removal between study and control group | Postoperatively in PACU from a minimum of 30 minutes till safe recovery from anaesthesia (approximately 1 hour)
  To compare the reliability of tragus pressure guided emergence from anaesthesia to conventional modes of recovery, studied by the timing and ease of removal of LMA.

CONTACTS AND LOCATIONS:
Overall Officials: Ashokka Balakrishnan, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhaskar SB. Emergence from anaesthesia: Have we got it all smoothened out? Indian J Anaesth. 2013 Jan;57(1):1-3. doi: 10.4103/0019-5049.108549. No abstract available. PMID 23716758
- [Background] Brown EN, Purdon PL, Van Dort CJ. General anesthesia and altered states of arousal: a systems neuroscience analysis. Annu Rev Neurosci. 2011;34:601-28. doi: 10.1146/annurev-neuro-060909-153200. PMID 21513454
- [Background] Academy of Medical Royal Colleges. Safe Sedation for Healthcare Procedures. Standards and Guidance. London: Academy of Medical Royal Colleges, 2013. http://www.aomrc.org.uk/doc_view/9737-safesedation- practice-for-healthcare-procedures-standards-and-guidance
- [Background] Buchanan FF, Myles PS, Cicuttini F. Effect of patient sex on general anaesthesia and recovery. Br J Anaesth. 2011 Jun;106(6):832-9. doi: 10.1093/bja/aer094. Epub 2011 May 9. PMID 21558068
- [Background] Checketts MR, Alladi R, Ferguson K, Gemmell L, Handy JM, Klein AA, Love NJ, Misra U, Morris C, Nathanson MH, Rodney GE, Verma R, Pandit JJ; Association of Anaesthetists of Great Britain and Ireland. Recommendations for standards of monitoring during anaesthesia and recovery 2015: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2016 Jan;71(1):85-93. doi: 10.1111/anae.13316. Epub 2015 Nov 19. PMID 26582586
- [Background] Lee B, Lee JR, Na S. Targeting smooth emergence: the effect site concentration of remifentanil for preventing cough during emergence during propofol-remifentanil anaesthesia for thyroid surgery. Br J Anaesth. 2009 Jun;102(6):775-8. doi: 10.1093/bja/aep090. Epub 2009 May 2. PMID 19411668
- [Background] Leslie K, Allen ML, Hessian EC, Peyton PJ, Kasza J, Courtney A, Dhar PA, Briedis J, Lee S, Beeton AR, Sayakkarage D, Palanivel S, Taylor JK, Haughton AJ, O'Kane CX. Safety of sedation for gastrointestinal endoscopy in a group of university-affiliated hospitals: a prospective cohort study. Br J Anaesth. 2017 Jan;118(1):90-99. doi: 10.1093/bja/aew393. PMID 28039246
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Pandit JJ, Cook TM. National Institute for Clinical Excellence guidance on measuring depth of anaesthesia: limitations of EEG-based technology. Br J Anaesth. 2013 Mar;110(3):325-8. doi: 10.1093/bja/aet006. No abstract available. PMID 23404965
- [Background] Punjasawadwong Y, Boonjeungmonkol N, Phongchiewboon A. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003843. doi: 10.1002/14651858.CD003843.pub2. PMID 17943802
- [Background] Singh R, Kharbanda M, Sood N, Mahajan V, Chatterji C. Comparative evaluation of incidence of emergence agitation and post-operative recovery profile in paediatric patients after isoflurane, sevoflurane and desflurane anaesthesia. Indian J Anaesth. 2012 Mar;56(2):156-61. doi: 10.4103/0019-5049.96325. PMID 22701207